CLINICAL TRIAL: NCT05241002
Title: The Application and Analysis of Diaphragm Electrical Impulse in Adult Patients With Spontaneous Breathing Trial: Before and After Tracheostomy
Brief Title: The Application and Analysis of Diaphragm Electrical Impulse in Adult Patients With Spontaneous Breathing Trial
Status: Terminated | Type: Observational
Why Stopped: Difficult to recruiting due to COVID-19 pandemic
Sponsor: Fu Jen Catholic University (Other)
Responsible Party: Principal Investigator, Ke-Yun, Chao, Leader of Respiratory Therapist, Fu Jen Catholic University
Other Study IDs: PL-2020100X
Record Dates: First submitted 2021-06-08; First posted 2022-02-15 (Actual); Last update posted 2022-10-27 (Actual); Status verified 2022-10

CONDITIONS: Tracheostomy
Keywords: tracheostomy; diaphragm electrical impulse; diaphragm activity; endotracheal tube

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of this study is to investigate the use of Edi in patients under the endotracheal tube and tracheostomy, and analysis of cardiopulmonary parameters in adult patients.

DETAILED DESCRIPTION:
Tracheostomy is a utilitarian surgical procedure of access; therefore, it should be discussed in light of the problem it addresses: access to the tracheobronchial tree. The trachea is a conduit between the upper airway and the lungs that delivers moist warm air and expels carbon dioxide and sputum. Failure or blockage at any point along that conduit can be most readily corrected with the provision of access for mechanical ventilators and suction equipment. In the case of upper airway obstruction, tracheostomy provides a path of low resistance for air exchange.

ELIGIBILITY:
Inclusion Criteria:

* Patents under planning tracheostomy will enroll to this study.

Exclusion Criteria:

* Pregnant women, age under 18 and unable to insert nasogastric tube

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patient in a single intensive care unit, under planning tracheostomy will enroll to this study.
Sampling Method: Probability Sample
Enrollment: 4 (Actual)
Dates: Start 2020-08-01 (Actual); Primary Completion 2022-03-31 (Actual); Study Completion 2022-04-30 (Actual)

PRIMARY OUTCOMES:
The electrical activity of the diaphragm (Edi) | one year
  Edi is the primary requirement for NAVA to function and the main source for ventilator trigger. This study will find the difference of data of Edi after surgery

SECONDARY OUTCOMES:
Cardiopulmonary function parameters | one year
  heart rate (HR)
Cardiopulmonary function parameters | one year
  blood pressure (BP)
Cardiopulmonary function parameters | one year
  stroke volume (SV)
Cardiopulmonary function parameters | one year
  cardiac output (CO)
Cardiopulmonary function parameters | one year
  total peripheral resistance (TPR)

CONTACTS AND LOCATIONS:
Locations (1):
- Fu Jen Catholic University Hospital, Fu Jen Catholic University, New Taipei City, Taiwan

REFERENCES:
- [Background] Demoule A, Jung B, Prodanovic H, Molinari N, Chanques G, Coirault C, Matecki S, Duguet A, Similowski T, Jaber S. Diaphragm dysfunction on admission to the intensive care unit. Prevalence, risk factors, and prognostic impact-a prospective study. Am J Respir Crit Care Med. 2013 Jul 15;188(2):213-9. doi: 10.1164/rccm.201209-1668OC. PMID 23641946
- [Background] Kallio M, Peltoniemi O, Anttila E, Jounio U, Pokka T, Kontiokari T. Electrical activity of the diaphragm during neurally adjusted ventilatory assist in pediatric patients. Pediatr Pulmonol. 2015 Sep;50(9):925-31. doi: 10.1002/ppul.23084. Epub 2014 Aug 7. PMID 25103680
- [Background] Goligher EC, Dres M, Fan E, Rubenfeld GD, Scales DC, Herridge MS, Vorona S, Sklar MC, Rittayamai N, Lanys A, Murray A, Brace D, Urrea C, Reid WD, Tomlinson G, Slutsky AS, Kavanagh BP, Brochard LJ, Ferguson ND. Mechanical Ventilation-induced Diaphragm Atrophy Strongly Impacts Clinical Outcomes. Am J Respir Crit Care Med. 2018 Jan 15;197(2):204-213. doi: 10.1164/rccm.201703-0536OC. PMID 28930478